CLINICAL TRIAL: NCT05323981
Title: A Single Center, Randomized, Double-blind, Parallel Controlled Phase I Trial Comparing the Pharmacokinetics and Safety of Two Specifications of HS627 Injection, a Recombinant Humanized Anti-Human Epidermal Growth Factor Receptor Monoclonal Antibody Injection, With PERJETA After a Single 420mg Intravenous Dose in Healthy Male Subjects
Brief Title: Comparison of Pharmacokinetics and Safety of HS627(2 Specifications) Versus PERJETA With a Single Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS627-TBE
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Similarity of Pharmacokinetics and Safety
MeSH Terms: interventions — pertuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HS627(210mg/7ml) (Experimental)
  Interventions: Drug: HS627(210mg/7ml)
- HS627(420mg/14ml) (Experimental)
  Interventions: Drug: HS627(420mg/14ml)
- PERJETA (Active Comparator)
  Interventions: Drug: Perjeta

INTERVENTIONS:
Drug: HS627(210mg/7ml) — Intravenous drip of 420mg HS627
  Arms: HS627(210mg/7ml)
Drug: HS627(420mg/14ml) — Intravenous drip of 420mg HS627
  Arms: HS627(420mg/14ml)
Drug: Perjeta — Intravenous drip of 420mg PERJETA
  Arms: PERJETA

SUMMARY:
To evaluate the bioequivalence of HS627(2 specifications) with PERJETA in a single intravenous administration in healthy subjects

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel controlled，single-dose phase I study to compare the pharmacokinetics and safety of HS627 (2 specifications) with PERJETA in Chinese healthy male adults

ELIGIBILITY:
Inclusion Criteria:

* 1. Signing the informed consent and being able to complete the test according to the plan;
* 2. Aged >= 18 and <= 40 (subject to the day of signing informed consent), male;
* 3. BMI is between 20~25 kg/m2 (including 20 kg/m2 and 25 kg/m2), and the weight is between 50-70kg (including 50kg and 70kg);
* 4. The left ventricular ejection fraction (LVEF) was more than 50% by echocardiography within 2 weeks before drug administration;
* 5. During the trial period and within 6 months after the infusion, the subjects or their spouses should take appropriate and effective contraceptive measures, such as abstinence and double barrier method (such as condom and diaphragm), oral contraceptive pill and IUD placement

Exclusion Criteria:

* 1. Patients with mental, respiratory, cardiovascular, digestive, urinary, reproductive, skeletal and motor diseases, blood, endocrine, nervous and other system diseases, and the judgment of the researchers has an impact on the pharmacokinetic results or safety;
* 2. Those who have a history of allergy to pertuzumab or any of its auxiliary materials or food; or who have a history of specific allergy (asthma, urticaria, eczema dermatitis, etc.); or who are allergic to the apparatus (such as syringe needle or intravenous drip needle, or intravenous drip hose) needed in the test;
* 3.Those who have special requirements for diet and cannot follow the unified diet;
* 4.Serious bleeding factors affecting peripheral venous blood collection;
* 5. Patients with history of malignancy;
* 6. Having previously received any antibody treatment targeting HER2 receptor or used monoclonal antibody within 6 months before signing informed consent;
* 7. Vaccinated with any live vaccine within 6 months before signing the informed consent;
* 8. Alcoholics or regular drinkers within 3 months before the test, i.e. those who drink more than 14 units of alcohol per week (14 bottles of 360 ml beer or 630 ml spirits with 40% alcohol or 2100 ml wine), or whose breath alcohol test is positive;
* 9. Have used soft drugs (such as marijuana) within 3 months before signing informed consent or hard drugs within 1 year before signing the informed consent (e.g. cocaine, phencyclidine, etc.); drug abuse test positive (morphine, Amphetamine, ketamine, dimethylene dioxoamphetamine, tetrahydrocannabinolic acid);
* 10. Within 3 months prior to signing the informed consent, he had blood donation history or lost more than 400ml of blood, received blood transfusion or had used blood products; those who lost more than 200 ml blood within one month before signing the informed consent;
* 11. Those who have participated in other clinical trials and used the experimental drugs or instruments within 3 months before signing the informed consent;
* 12. Those who are addicted to smoking or have more than 5 cigarettes per day on average within three months before signing the informed consent;
* 13. Those who have undergone surgery within 2 months before signing the informed consent;
* 14. Those who have received any drug treatment (including prescription drugs, over-the-counter drugs, biological products, proprietary Chinese medicine, vitamins, dietary supplements, etc.) and health care products within 14 days prior to signing the informed consent, or whose previous treatment drug(s) is(are) still within 5 half-lives when using the experimental drugs;
* 15. Patients with upper respiratory tract infection or other acute infections within 2 weeks before screening;
* 16. Drinking too much tea, coffee and / or caffeinated drinks (more than 8 cups, 1 cup = 250 ml) every day;
* 17. In screening or baseline period, the researchers judge that the vital signs, physical examination and laboratory examination were abnormal with clinical significance;
* 18. In screening period or baseline period, the investigator judges the ECG be clinically significantly abnormal, or QTc >= 450 ms, or with a history of clinically significant ECG abnormalities;
* 19. Any positive result of HIV antibody, HBsAg, HCV antibody and Treponema pallidum antibody;
* 20. Anti-drug antibody (ADA) test is positive;
* 21. The researcher thinks whoever is not suitable to join the group or may not be able to complete the trial due to other reasons;
* 22. Researchers, staff of research centers, sponsors and employees or related personnel of contract research organizations.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-10-09 (Actual)

PRIMARY OUTCOMES:
（AUC0-∞）of HS627(2 specifications) and PERJETA | 85Days
  Area under the concentration-time curve (AUC0 - ∞) from 0 to infinity of HS627(2 specifications) and PERJETA

SECONDARY OUTCOMES:
（AUC0-t）of HS627(2 specifications) and PERJETA | 85Days
  Area under the concentration-time curve (AUC0 - ∞) from 0 to the last measurable concentration of HS627(2 specifications) and PERJETA
Cmax | 85Days
  The maximal concentration of HS627 (2 specifications) and PERJETA
Tmax | 85Days
  The timepoint at which Cmax reached
CL | 85Days
  Rate of plasma drug clearance
T1/2 | 85Days
  Half life
Vd | 85Days
  Volume of distribution of HS627 (2 specifications) and PERJETA

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China